CLINICAL TRIAL: NCT02394223
Title: Full Field Optical Coherence Tomography of Prostate Biopsies for the Diagnosis of Prostate Cancer
Brief Title: FFOCT for the Diagnosis of Prostate Cancer
Acronym: BIOMAGIC01
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOK 13142
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Patients With PSA Level 4.0 ng/mL
Keywords: Cancer; Prostate; PSA; Biopsies; FFOCT procedure
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Full Field Optical Coherence Tomography (FFOCT) procedure
  Interventions: Procedure: Full Field Optical Coherence Tomography (FFOCT) procedure

INTERVENTIONS:
Procedure: Full Field Optical Coherence Tomography (FFOCT) procedure — TRUS Prostate biopsy are performed under the care procedure Pathological examination of these prostate biopsy with FFOCT procedure, as compared to standard pathological evaluation

SUMMARY:
Primary objective :

The primary objective is to evaluate the diagnosis performance of FFOCT for cancer detection in patients undergoing TRUS prostate biopsy, as compared to standard pathological evaluation.

Secondary objective:

* Evaluate predictive values of FFOCT for cancer detection on prostate biopsy cores
* Evaluate the value of FFOCT for cancer characterization on prostate biopsy cores
* Evaluate the reproducibility of FFOCT evaluation for cancer detection on prostate biopsy cores
* Evaluate the learning curve of FFOCT evaluation on prostate biopsy cores
* Evaluate FFOCT procedure time

DETAILED DESCRIPTION:
Research in optical imaging has led to the development of the Full Field Optical Coherence Tomography (FFOCT) technology, which allows to image fresh tissues up to a depth of a few hundreds microns. The system is a microscope coupled with an interferometer. A halogen light source is used to illuminate the tissue specimen and a reference mirror. The light retro diffused by the specimen is combined with the light reflected by the mirror, and the interference signal is measured. Multiple Grey scale images are obtained and automatically stitched to obtain a complete slide throughout the specimen. The feasibility of the technique has been reported in various pilot studies, as well as the absence of any potential tissue harm and subsequent pathological artifact caused by the process.

FFOCT could be used as an additional detection tool for prostate cancer screening. The use of extended systematic trans-rectal ultrasound-guided (TRUS) prostate biopsies has led to over-diagnosis and over-treatment. Also, the number of unnecessary biopsies has increased, along with the morbidity of the procedure. Performing a "pre-pathological" evaluation of biopsy cores during the biopsy procedure would be of significant help to determine the nature of targeted areas and guide the number of biopsies to perform.

We hypothesize that FFOCT imaging of prostate biopsy cores would allow a cancer detection rate not statistically different from pathological analysis.

ELIGIBILITY:
Inclusion Criteria:

* - Patient aged 45 to 75 years old included
* - PSA level 4.0 ng/mL
* - Patient referred for trans rectal ultrasound-guided prostate biopsy with additional MRI-targeted biopsies
* - Patient no opposed to participate in the study
* Patient affiliated to the French National Social Security System

Exclusion Criteria:

* Known prostate cancer
* Patients unable to understand the course of the study

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 45 to 75 years old, with PSA level 4.0 ng/mL
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2016-01-27 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2017-01-27 (Actual)

PRIMARY OUTCOMES:
To evaluate the diagnosis performance of FFOCT for cancer detection in patients undergoing TRUS prostate biopsy, as compared to standard pathological evaluation | One day (biopsy procedure)
  Presence or absence of prostate cancer on pathological examination of prostate biopsy cores

SECONDARY OUTCOMES:
To evaluate the predictive values of FFOCT for cancer detection on prostate TRUS biopsy | One day (biopsy procedure)
  the positive and negative predictive values for the presence of cancer, based on the prevalence of cancer in the population studied
To evaluate the value of FFOCT for cancer characterization on prostate biopsy cores | One day (biopsy procedure)
  Gleason score and cancer length of prostate cancer on pathological examination of each prostate biopsy cores
To evaluate the reproducibility of FFOCT evaluation for cancer detection on prostate biopsy cores | One day (biopsy procedure)
  the inter observer agreement for the diagnosis of cancer between 2 experienced pathologists fully trained to the technique, as well as 2 experienced urologists trained to the technique
To evaluate the learning curve of FFOCT evaluation on prostate biopsy cores | One day (biopsy procedure)
  the evolution of the diagnostic performance with time when FFOCT images are evaluated with an experienced pathologist untrained to the technique before the beginning of the study
To evaluate FFOCT procedure time | One day (biopsy procedure)
  the duration of FFOCT procedure

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Barry Delongchamps, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance Publique - Hôpitaux de Paris Cochin Hospital, Paris, France